CLINICAL TRIAL: NCT06963658
Title: Acute Effect of Isometric Excercise on Pain Sensitivity in Adults With Chronic Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taif University (Other)
Responsible Party: Principal Investigator, Hosam Alzahrani, Associate professor, Taif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISO-Ex 0011112222
Record Dates: First submitted 2025-03-13; First posted 2025-05-09 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Chronic Low Back Pain (CLBP)
Keywords: pain sensitivity; isometric exercise; low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multiple repetition isometric wall squat (Experimental): Participants were directed to rest their backs against the wall with shoulder width apart and feet parallel, then descend until they achieve an angle of 100 degrees at knee joint. The knee joint angle was assessed using a goniometer placed on the lateral epicondyle of the knee, aligned with the femur, while the anchor arm was aligned with the lateral malleolus. They were instructed to maintain the isometric hold for up to three minutes, or until volitional fatigue was reached.with a 30-second rest period between each squat hold.
  Interventions: Other: Multiple repetition isometric wall squat
- Multiple Isometric wall squat exercise + Double Leg Lower with Isometric Hold (Experimental): Participants were directed to rest their backs against the wall with shoulder width apart and feet parallel, then descend until they achieve an angle of 100 degrees at knee joint. The knee joint angle was assessed using a goniometer placed on the lateral epicondyle of the knee, aligned with the femur, while the anchor arm was aligned with the lateral malleolus. They were instructed to maintain the isometric hold for up to three minutes, or until volitional fatigue was reached.with a 30-second rest period between each squat hold.
  Immediately post 60 second rest, Determine the participant's maximum angle using the double leg lowering test from supine position let the participant with both legs straightened before lifting the posterior hip, lowering the legs to a specific angle. Turn on the stopwatch. Hold the position near--maximally, try to achieve on (IES=9/10) and hold for the longest duration. They should reach 4 minutes for 3 repetition with 30 seconds rest between repetition
  Interventions: Other: Multiple Isometric wall squat exercise + Double Leg Lower with Isometric Hold
- Control quiet seated rest (Experimental): The CON group served as the control group and did not perform any exercise. Participants were instructed to sit quietly in a standard height stationary clinical room patient chair for the entire eight minutes.
  Interventions: Other: Control quiet seated rest

INTERVENTIONS:
Other: Multiple repetition isometric wall squat — Participants were directed to rest their backs against the wall with shoulder width apart and feet parallel, then descend until they achieve an angle of 100 degrees at knee joint. The knee joint angle was assessed using a goniometer placed on the lateral epicondyle of the knee, aligned with the femur, while the anchor arm was aligned with the lateral malleolus. They were instructed to maintain the isometric hold for up to three minutes, or until volitional fatigue was reached.with a 30-second rest period between each squat hold.
  Arms: Multiple repetition isometric wall squat
Other: Multiple Isometric wall squat exercise + Double Leg Lower with Isometric Hold — Participants were directed to rest their backs against the wall with shoulder width apart and feet parallel, then descend until they achieve an angle of 100 degrees at knee joint. The knee joint angle was assessed using a goniometer placed on the lateral epicondyle of the knee, aligned with the femur, while the anchor arm was aligned with the lateral malleolus. They were instructed to maintain the isometric hold for up to three minutes, or until volitional fatigue was reached.with a 30-second rest period between each squat hold. Immediately post 60 second rest, Determine the participant's maximum angle using the double leg lowering test from supine position let the participant with both legs straightened before lifting the posterior hip, lowering the legs to a specific angle. Turn on the stopwatch. Hold the position near--maximally, try to achieve on (IES=9/10) and hold for the longest duration. They should reach 4 minutes for 3 repetition with 30 seconds rest between repetition
  Arms: Multiple Isometric wall squat exercise + Double Leg Lower with Isometric Hold
Other: Control quiet seated rest — The control group served as the control group and did not perform any exercise. Participants were instructed to sit quietly in a standard height stationary clinical room patient chair for the entire eight minutes.
  Arms: Control quiet seated rest

SUMMARY:
Randomized control trial to examine the immediate effect of isometric exercise on pressure pain threshold (PPT) in adults with chronic low back pain. The secondary aim of this study was to investigate the acute effects of isometric exercise on clinical pain intensity.

DETAILED DESCRIPTION:
Participants will attend a single visit to the hospital for two hours, which will include collecting demographic details and clinical characteristics through self-reported assessment scales. After that, outcome measures (pain sensitivity and current low back pain intensity) were collected prior to the intervention and repeated immediately post-intervention.

ELIGIBILITY:
Inclusion Criteria :

1. participants aged ≥18 years or older
2. participant diagnosed with non-specific chronic lower back pain (> 12 weeks)
3. Able to perform physical therapy excercise . Exclusion criteria : The study will exclude

1- pregnant women 2- lactating women for one or less than one year post-natal. 3- any certain medical conditions that could interfere with physical activity, including:

* uncontrolled diabetes
* cardiovascular problem
* orthopedic impairments
* balance problems. 4-serious spinal pathologies :
* infection
* fractures
* tumors
* inflammatory diseases like ankylosing spondylitis 5- neurological compromise,
* spinal nerve compromise
* cauda equina syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is pain sensitivity | pre- and immediately post-intervention
  Pain sensitivity was assessed via pressure pain threshold (PPT) using a standard procedure. The PPT was assessed by a digital pressure algometer (Wagner digital force Ten FDX 25 with 1 cm 2 rubber tip).This instrument has been widely utilized in various studies and has been shown to be valid and reliable in assessing PPT among people with musculoskeletal pain. If post intervention PPT was higher than pre-intervention value, this indicated that pain sensitivity decreased, suggesting exercise induced hypoalgesia occurred. If post-intervention PPT was lower than pre-intervention PPT, this indicates that pain sensitivity increased, suggesting that exercise induced hyperalgesia occurred.

SECONDARY OUTCOMES:
The secondary outcome is the pain intensity in the lower back | pre- and immediately post-intervention
  It is a subjective rating of pain intensity in the lower back using a visual analog scale,where a rating of zero indicates that participant don't have pain and a rating of 10 indicates that the most severe pain. The VAS is reliable and valid for measuring pain in individuals with chronic musculoskeletal conditions. A change of one point in pain intensity on this scale is regarded as the minimal clinically important difference.

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdullah Hospital in bisha, Bisha, 'Asir Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No